CLINICAL TRIAL: NCT02021604
Title: The Use of Fluorodopa F 18 Positron Emission Tomography Combined With Computed Tomography in Congenital Hyperinsulinism and Insulinoma
Brief Title: Fluorodopa F 18 in Congenital Hyperinsulinism and Insulinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cook Children's Health Care System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-060
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Congenital Hyperinsulinism; Insulinoma
Keywords: Congenital Hyperinsulinism; HI; Hypoglycemia; FDOPA; 18F-DOPA; Hyperinsulinism; Insulinoma
MeSH Terms: conditions — Congenital Hyperinsulinism; Insulinoma; Hypoglycemia; Hyperinsulinism | interventions — fluorodopa F 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pancreatic Imaging with Fluorodopa F 18 (Experimental)
  Interventions: Drug: Fluorodopa F 18

INTERVENTIONS:
Drug: Fluorodopa F 18 — A dose of Fluorodopa F 18, 3-6 MBq/Kg (0.08-0.16 mCi/kg), will be injected intravenously into the subject under the direct supervision of the radiology sub-investigator. Then, the PET imaging procedure will begin and proceed for up to 70 minutes after injection. An abdominal CT image will be made using intravenous contrast. Both images, PET and CT, will be co-localized by the radiologist for interpretation.
  Other Names: Fluorodopa 18F (International Non-Proprietary Name); 6-[18F]fluorolevodopa (U.S. Pharmacopeia); Fluorodopa F 18 (CAS Number 75290-51-6)

SUMMARY:
Low blood sugars are known to cause brain damage in newborn babies. One of the most common causes of low blood sugars persisting beyond the new born period is a condition called congenital hyperinsulinism (HI). This is a disease whereby the pancreas secretes too much insulin and causes low blood sugars. Twenty to forty percent of these babies will have brain damage. There are two forms of this disease. In one form only a small part of the pancreas makes too much insulin (focal HI) and in the other, the whole pancreas make too much insulin (diffuse HI). Another very similar disease is insulinoma which occurs after birth, but also causes hyperinsulinism. If a surgeon could know which part of the pancreas has the focal lesion he could remove it and cure the patient.

The purpose of this study is to investigate whether a new investigational drug called Fluorodopa F 18, when used with a PET scan, can find the focal lesion and guide the surgeon to remove it, thus curing the patient and preventing further brain damage.

DETAILED DESCRIPTION:
Congenital Hyperinsulinism (HI) is a disorder of insulin secretion that causes profound hypoglycemia leading to significant morbidity. It is the most common form of persistent neonatal hypoglycemia, and the most dangerous. Inappropriate insulin secretion causes not only hypoglycemia but also inability to release free fatty acids from adipose tissue and inability to release glycogen from the liver. Hence the brain is deprived of all the major fuel sources (glucose, beta-hydroxybutyrate and lactate) for energy thus leading to the high incidence of brain damage. In up to 50% of cases of congenital hyperinsulinism, medical therapy fails and surgical resection of the pancreas is necessary. Previous techniques developed to differentiate those patients with focal HI in whom surgery could result in a cure are very invasive and put the infants at risk for hypoglycemic brain damage or arterial thrombosis.

It is known that the beta cells in the pancreatic islets, similar to other neuroendocrine tissues, contain amino acid decarboxylase (AADC). Beta cells take up L-Dopa and convert it into dopamine by AADC. It was proposed that as other neuroendocrine tumors such as phaeochromocytoma and carcinoid tumors express AADC and can be very easily visualized using Fluorodopa F 18 PET then so also would the pancreas be easily and accurately visualized. After initial reports demonstrated the effectiveness, safety and accuracy, there have been now over 200 patients with HI reported in the literature who have had Fluorodopa F 18 PET scans with suggestions that referral to major HI centers for Fluorodopa F 18 PET CT is now an integral part of standard of care management of patients with HI that require surgery. Fluorodopa F 18 PET scanning for patients with Hyperinsulinism is now established in Europe and Australia, and has close to 95% sensitivity. When linked to Computed Tomography (CT) image of the pancreas, Fluorodopa F 18 PET allows the surgeon to image the pancreas in three dimensions, to even more accurately identify the site of the focal lesion, increasing the chance of a sufficient partial pancreatectomy to cure the patient.

Similarly, insulinomas are neuroendocrine cell tumors that are typically benign (90%) and very rare occurring in 1-4 per million of the population with > 50% occurring in adults >age 25 years. Biochemical differentiation of insulinomas from congenital hyperinsulinism may be aided by the use of the pro-insulin:insulin ratio, by the age of presentation and by the history. The standard of care for insulinoma is to remove them once identified, rather than long term medical treatment. Current imaging techniques include CT scan pancreas, endoscopic ultrasound of the pancreas and MRI pancreas however despite using these modalities in some patients the insulinoma may not be found. 18F-DOPA has been shown to be superior than MIBG scanning for neuroendocrine tumors such as phaeochromocytoma, but there is very little data in patients with insulinoma. Moreover, patients with MEN 1 and insulinoma may have more than one tumor, which if missed with conventional imaging could result in failure to cure with surgery.

The objectives of this study are:

1. To determine, using Positron Emission Tomography, whether or not the uptake of a radiopharmaceutical agent, Fluorodopa 18F (18F-DOPA) produced in a cyclotron located at a distance far from the imaging center will produce qualitatively adequate pancreatic images in patients with congenital hyperinsulinism
2. To determine, using direct comparisons, whether or not Fluorodopa 18F Positron Emission Tomography (18F-DOPA PET) combined with Computed Tomography (CT) will produce pancreatic images matching the gold-standard of histopathological findings at surgery for partial or complete pancreatectomy in the treatment of patients with congenital hyperinsulinism
3. To determine, using direct comparisons, whether or not Fluorodopa 18F Positron Emission Tomography (18F-DOPA PET) combined with Computed Tomography (CT) will produce pancreatic images matching the gold-standard of histopathological findings at surgery for insulinomas
4. To determine the best way to interpret the 18F-DOPA PET scans comparing SUV max:SUV sub max at a ratio of the current 1.5, a suggested 1.3 and by using visual inspection of the images.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HI attending the Cook Children's Congenital Hyperinsulinism Center and being treated by an Endocrinologist which may be the PI or a partner of this clinician.
* The patient's Endocrinologist has determined that the patient cannot be safely managed with standard medical therapy (failed) and surgery is recommended to prevent future episodes of severe hypoglycemia and preserve brain function. Failure of medical therapy is defined as both:

  * Hypoglycemia (blood glucose <70 m/dL) on a single measure despite the use of anti-hypoglycemic medications, if applicable to the individual patient, including and limited to diazoxide or octreotide
  * Inability to fast, defined as the inability to maintain a blood glucose >50 mg/dL for: 1) more than 12 hours for infants < 1 year of age; 2) more than 15 hours 1-3 years of age; 3) more than 18 hours over 3 years of age
* Patients in whom the genetic testing (if available and informative) does not prove diffuse HI disease. Such children might be considered if they have one or more of the following situations:

  * no genetic testing results (e.g., due to insurance denial or parental refusal)
  * negative genetic testing (note: only 75% of mutations may be found with existing technology)
  * no autosomal recessive mutations in ABCC8 or KCNJ11 on the maternal allele
  * no autosomal dominant mutations in ABCC8 or KCNJ11
* Patients thought to have focal HI disease based on genetic testing or insulinoma based on clinical evaluation and have well-controlled blood glucose levels with any degree of dietary or medical management, BUT the patient and their parent(s) or LAR wishes to proceed with surgery for a possible cure of HI disease.

Exclusion Criteria:

* Patients who do not have a diagnosis of HI
* Patients with genetic evidence of diffuse HI
* Patients who are pregnant
* Nursing mothers who are unwilling to discontinue breastfeeding their infant for 48 hours after Fluorodopa F 18 injection
* Patients with a known allergy to Fluorodopa F 18 agent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-10-09 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Radioactivity of 18F-DOPA following transport | 1 day
  Positron Emission Tomography will be used to determine whether or not the uptake of a radiopharmaceutical agent, Fluorodopa F 18, produced in a cyclotron located at a distance far from the imaging center will produce qualitatively adequate pancreatic images in patients with congenital hyperinsulinism
Accuracy of PET imaging compared to intraoperative pancreatic biopsy in patients with congenital hyperinsulinism | up to one month
  Investigators will directly compare pancreatic images from Fluorodopa F 18 PET combined with Computed Tomography versus the gold-standard of histopathological findings at surgery in subjects who received a partial or complete pancreatectomy

SECONDARY OUTCOMES:
Accuracy of PET imaging compared to intraoperative pancreatic biopsy in patients with insulinoma | up to one month
  Investigators will directly compare pancreatic images from Fluorodopa F 18 PET combined with Computed Tomography versus the gold-standard of histopathological findings at surgery in subjects who received a partial or complete pancreatectomy
Ratio of Standard Uptake Value max to sub max | up to one month
  Investigators will compare SUV max to SUV sub max at a ratio of the current 1.5, a suggested 1.3 and by using visual inspection of the images.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Thornton, MD, Principal Investigator — Cook Children's Health Care System
Locations (1):
- Cook Children's Medical Center, Fort Worth, Texas, United States

REFERENCES:
- [Background] de Lonlay-Debeney P, Poggi-Travert F, Fournet JC, Sempoux C, Dionisi Vici C, Brunelle F, Touati G, Rahier J, Junien C, Nihoul-Fekete C, Robert JJ, Saudubray JM. Clinical features of 52 neonates with hyperinsulinism. N Engl J Med. 1999 Apr 15;340(15):1169-75. doi: 10.1056/NEJM199904153401505. PMID 10202168
- [Background] Thornton PS, Finegold DN, Stanley CA, Sperling MA. Hypoglycemia in the infant and child. In Sperling MA ed. Pediatric Endocrinology 2nd ed., pp 367-84. Philadelphia: Saunders, 2002.
- [Background] Stanley CA, Thornton PS, Finegold DN, Sperling MA: Hypoglycemia in neonates and infants. In Sperling MA ed. Pediatric Endocrinology 2nd edition chpt 7 pages 135-59. 2002.
- [Background] Suchi M, Thornton PS, Adzick NS, MacMullen C, Ganguly A, Stanley CA, Ruchelli ED. Congenital hyperinsulinism: intraoperative biopsy interpretation can direct the extent of pancreatectomy. Am J Surg Pathol. 2004 Oct;28(10):1326-35. doi: 10.1097/01.pas.0000138000.61897.32. PMID 15371948
- [Background] Jager PL, Chirakal R, Marriott CJ, Brouwers AH, Koopmans KP, Gulenchyn KY. 6-L-18F-fluorodihydroxyphenylalanine PET in neuroendocrine tumors: basic aspects and emerging clinical applications. J Nucl Med. 2008 Apr;49(4):573-86. doi: 10.2967/jnumed.107.045708. Epub 2008 Mar 14. PMID 18344441
- [Background] Otonkoski T, Nanto-Salonen K, Seppanen M, Veijola R, Huopio H, Hussain K, Tapanainen P, Eskola O, Parkkola R, Ekstrom K, Guiot Y, Rahier J, Laakso M, Rintala R, Nuutila P, Minn H. Noninvasive diagnosis of focal hyperinsulinism of infancy with [18F]-DOPA positron emission tomography. Diabetes. 2006 Jan;55(1):13-8. PMID 16380471
- [Background] Mohnike K, Blankenstein O, Minn H, Mohnike W, Fuchtner F, Otonkoski T. [18F]-DOPA positron emission tomography for preoperative localization in congenital hyperinsulinism. Horm Res. 2008;70(2):65-72. doi: 10.1159/000137655. Epub 2008 Jun 12. PMID 18547951
- [Background] Hardy OT, Hernandez-Pampaloni M, Saffer JR, Suchi M, Ruchelli E, Zhuang H, Ganguly A, Freifelder R, Adzick NS, Alavi A, Stanley CA. Diagnosis and localization of focal congenital hyperinsulinism by 18F-fluorodopa PET scan. J Pediatr. 2007 Feb;150(2):140-5. doi: 10.1016/j.jpeds.2006.08.028. PMID 17236890
- [Background] Hardy OT, Hernandez-Pampaloni M, Saffer JR, Scheuermann JS, Ernst LM, Freifelder R, Zhuang H, MacMullen C, Becker S, Adzick NS, Divgi C, Alavi A, Stanley CA. Accuracy of [18F]fluorodopa positron emission tomography for diagnosing and localizing focal congenital hyperinsulinism. J Clin Endocrinol Metab. 2007 Dec;92(12):4706-11. doi: 10.1210/jc.2007-1637. Epub 2007 Sep 25. PMID 17895314
- See also: Cook Children's Endocrinology — http://www.cookchildrens.org/endocrinology/Pages/default.aspx